CLINICAL TRIAL: NCT06899854
Title: Collection of Blood and Tissue Samples From Patients With Primary Liver Cancer Undergoing Systemic Therapy, Surgical Resection, or Liver Biopsy.
Brief Title: Collection of Blood and Tissue Samples From Patients With Primary Liver Cancer.
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Mario Mondelli, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: p_129_2023
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC); Cholangiocarcinoma
Keywords: immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with HCC: Patients with a diagnosis of HCC
- Patients with CCA: Patients with a diagnosis of CCA

SUMMARY:
The project aims to collect blood, tissue samples, and clinical data from patients with primary liver cancer (mainly hepatocellular carcinoma and intrahepatic cholangiocarcinoma) undergoing systemic therapy, surgical resection, or liver biopsy. Primary liver cancer is a growing global health challenge, with over one million cases expected by 2025 and a lack of effective treatments. The three-year study will systematically collect and store samples to support translational research for new therapies. Blood will be drawn at key points during systemic therapy, while tissue samples will be obtained from surgical resections or biopsies, provided they are not needed for diagnostics.

DETAILED DESCRIPTION:
The project aims to collect blood and tissue samples, as well as clinical data, from patients with primary liver cancer undergoing systemic therapy, surgical resection, or liver biopsy.

Primary liver cancers represent a global health challenge, with an estimated incidence exceeding one million cases by 2025. Hepatocellular carcinoma (HCC) is the most common form, accounting for approximately 90% of cases. The second most common type, intrahepatic cholangiocarcinoma (iCCA), is an epithelial tumor arising along second-order bile ducts, often in patients without known risk factors.

The lack of effective therapies, along with the increasing incidence and mortality rates, drives the need to explore new therapeutic approaches. These approaches require robust translational studies, which can only be conducted through the systematic collection of biological samples from patients undergoing systemic therapy.

The three-year study plans to collect, process, and store blood and tissue samples from patients with primary liver cancer undergoing systemic therapy, surgical resection, or liver biopsy.

For each patient undergoing systemic therapy, blood will be drawn at the start of therapy, during clinical follow-ups (first three), at the end of therapy, and at the first post-therapy imaging assessment. From patients undergoing surgical resection, in addition to blood, a tissue sample not required for diagnostic purposes will be obtained. If a patient undergoes a liver biopsy and consents to participate in the study, a blood sample will be collected, and a biopsy tissue sample not needed for diagnostic purposes will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Primary liver cancer (hepatocellular carcinoma or intrahepatic cholangiocarcinoma)

Signed informed consent

Patient eligible to start first-line systemic therapy

Patient eligible for surgical resection

Exclusion Criteria:

Concurrent conditions with a life expectancy of less than 12 months

Autoimmune or chronic inflammatory diseases

Substance abuse dependency

Other active extrahepatic malignancies or those treated within the last 3 years, except for the following exceptions:

Tumors resected with curative intent and with no evidence of disease recurrence for >3 years prior to signing the informed consent, considered at low risk of recurrence

Adequately resected non-melanoma skin cancers or lentigo maligna with no evidence of metastasis

Adequately treated carcinoma in situ of the cervix with no evidence of recurrence

Prostatic intraepithelial neoplasia with no evidence of infiltrative disease

Adequately treated non-invasive papillary urothelial tumors or urothelial carcinoma in situ

HIV infection

Lack of patient cooperation or failure to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of HCC or CCA eligible to start first-line systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with HCC or CCA as assessed by extraction of PBMC and infiltrating cells | From enrollment to the end of treatment at 6 months
  The primary objective of the study is the collection of peripheral blood samples to extract mononuclear cells and serum, as well as tissue samples to extract infiltrating cells and tumor cells. As regards the peripheral blood the extraction will be performed by Ficoll stratification. Infiltrating cells in the tissue will be isolated by enzymatic and mechanical dissociation of the tissue and centrifugation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided